CLINICAL TRIAL: NCT03633682
Title: Evaluation of Text Message Engagement Support of Mindfulness Smartphone
Brief Title: Evaluation of Text Message Engagement Support of Mindfulness Smartphone Applications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Stephen Schueller, Adjunct Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00206204
Record Dates: First submitted 2018-06-26; First posted 2018-08-16 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Engagement Support (Experimental): In the engagement support group, participants will be sent text messages that will encourage use of the app through tips, reminders, and encouraging messages.
  Interventions: Behavioral: Headspace - Meditation and Mindfulness App; Behavioral: Stop, Breathe, & Think - Meditation and Mindfulness App
- No Engagement Support (Other): Participants in this group will receive no text message support.
  Interventions: Behavioral: Headspace - Meditation and Mindfulness App; Behavioral: Stop, Breathe, & Think - Meditation and Mindfulness App

INTERVENTIONS:
Behavioral: Headspace - Meditation and Mindfulness App — Participants randomized to this arm will receive 1-month full access to the Headspace meditation app. They will be asked to listen to at least one meditation a day over the four week study period. Mindfulness is the ability to intentionally and nonjudgementally observe thoughts, bodily sensations, or feelings in the present moment. The apps include guided mindfulness meditations targeting several different areas, such as stress, anxiety, compassion, and sleep.
Behavioral: Stop, Breathe, & Think - Meditation and Mindfulness App — Participants randomized to this arm will receive 1-month full access to the Stop, Breathe, & Think meditation app. They will be asked to listen to at least one meditation a day over the four week study period. Mindfulness is the ability to intentionally and nonjudgementally observe thoughts, bodily sensations, or feelings in the present moment. The apps include guided mindfulness meditations targeting several different areas, such as stress, anxiety, compassion, and sleep.

SUMMARY:
The aim of this study is to assess the usability of two mindfulness smartphone applications (apps) and to evaluate whether text message support can promote engagement with those apps through a 4-week trial comparing support vs. no support.

DETAILED DESCRIPTION:
Part one of this study is to conduct usability testing to understand more about the acceptability and usability of these existing mindfulness apps in a population with depression and anxiety. The goal of usability testing is to identify any usability problems, provide information for future app development, and determine the participant's satisfaction with the apps. Participants will then be randomized to receive either engagement support or no support which will be delivered via text messaging, and will be randomized to use one of the two mindfulness applications for the 4 week period. Specific Aim 2.1 is to evaluate any differences on outcome measures between the two mindfulness apps. Specific Aim 2.2 is to evaluate the differences of outcome measures between text message engagement support versus no support, regardless of the mindfulness app. For Aim 2.1, the investigators predict that all mindfulness apps will be capable of leading to improvements on outcome measures. For Aim 2.2, the investigators predict that the text message engagement support arm will engage more with the mindfulness app and will see greater improvements in outcome measures regardless of the mindfulness app.

ELIGIBILITY:
Inclusion Criteria:

1. meet criteria for clinically significant distress caused by anxiety defined by a Generalized Anxiety Disorder-7 (GAD-7) greater than a 10 or clinically significant distress caused my depression defined by a Patient Health Questionnaire (PHQ-9) greater than 10
2. 18 years of age or older;
3. fluent in English;
4. lives in the Chicago area and are able to attend and in person session;
5. own an internet ready smartphone with data and text plans.

Exclusion Criteria:

1. have visual, hearing, voice, or motor impairment that would prevent completion treatment procedures;
2. past or current diagnosis of a psychotic disorder, bipolar disorder, dissociative disorder, substance or alcohol abuse dependence, or other diagnosis for which participation in the trial would be dangerous;
3. suicidal, defined as a 1 or higher on item 9 of the Patient Health Questionnaire (PHQ-9);
4. adults unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Depression and Anxiety at Week 2 and Week 4 | Baseline, Week 2, Week 4
  Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item self-report measure of depression. Scores on this measure range from 0 (Not At All) to 3 (Nearly Every Day).
Change in Anxiety at Week 2 and Week 4 | Baseline, Week 2, Week 4
  Generalized Anxiety Disorder 7-item scale (GAD-7). The GAD-7 is a 7-item self-report measure of anxiety. Scores on this measure range from 0 (Not At All) to 3 (Nearly Every Day).

SECONDARY OUTCOMES:
App Usage | Week 1, Week 2, Week 3, Week 4
  App usage will be defined as how many minutes the participant meditated and how many meditations they listened to.
App Satisfaction | Week 1, Week 2, Week 3, Week 4
  App satisfaction evaluates the participants satisfaction with the app on a scale ranging from 1 (Not At All) to 5 (Extremely).

OTHER OUTCOMES:
Change in Mindfulness at Week 4 | Baseline and Week 4
  Five Facet Mindfulness Questionnaire. A self-report measure of five facets of mindfulness: observing, describing, acting with awareness, being nonjudgmental, and nonreactivity. The FFMQ is a 39-item questionnaire, and each FFMQ item is rated on a 5-point scale ranging from 1 ("never or very rarely true") to 5 ("very often or always true").
Change in Psychological Flexibility at Week 2 and Week 4 | Baseline, Week 2, Week 4
  Acceptance and Action Questionnaire (AAQ-II). The AAQ-II is a 7-item self-report questionnaire designed to measure psychological flexibility. Scores on this measure range from 1 (never true) to 7 (always true).
Change in Depression, Anxiety, and Stress at Week 1, 2, 3, and 4 | Baseline, Week 1, Week 2, Week 3, Week 4
  Depression, Anxiety, and Stress Scale (DASS). The DASS-21 is a 21-item self-report measure consisting of three subscales (depression, anxiety and stress). Answers range from 0 (did not apply to me at all) to 3 (applied to me very much).
Change in Rumination at Week 4 | Baseline, Week 4
  The Rumination-Reflection Questionnaire (RRQ). The RRQ is a 24-item self-reported questionnaire assessing both self-rumination and self-reflection, with 12 items corresponding to each subscale. Participants rate the degree to which they engage in self- rumination (e.g. "sometimes it is hard for me to shut off thoughts about myself") and self-reflective thoughts (e.g. "I love to meditate on the nature and meaning of things") on a Likert scale ranging from one (strongly disagree) to five (strongly agree).
Change in Insomnia at Week 4 | Baseline, Week 4
  Insomnia Severity Scale (ISI). The ISI is a 7-item self-report measure of insomnia. Total ISI scale scores range from a low of 0 (least insomnia) to a high of 28 (worst insomnia)
Change in Quality of Life at Week 4 | Baseline, Week 4
  Quality of Life Scale (QOLS). The QOLS is a 16-item self-report measure of quality of life. The QOLS accesses five conceptual domains of quality of life: material and physical well-being, relationships with other people, social, community and civic activities, personal development and fulfillment, and recreation. The scale ranges from 1 (terrible) to 7 (delighted).
Change in Stress at Week 4 | Baseline, Week 4
  Perceived Stress Scale (PSS). The PSS is a 10-item self-report measure of stress, with scores ranging from 10-40 and a higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwester University, Feinberg School of Medicine, Center for Behavioral Intervention Technologies, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

DOCUMENTS (2):
  • Study Protocol (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT03633682/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT03633682/SAP_002.pdf